CLINICAL TRIAL: NCT00406419
Title: A Randomized, Double-Blind, Parallel Group, International Study to Evaluate the Safety and Efficacy of Ocrelizumab Compared to Placebo in Patients With Active Rheumatoid Arthritis Continuing Methotrexate Treatment
Brief Title: A Study of Ocrelizumab Compared to Placebo in Patients With Active Rheumatoid Arthritis Continuing Methotrexate Treatment (STAGE)
Acronym: STAGE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on analysis of results and consideration of available treatments, the overall benefit to risk profile of ocrelizumab was not favorable in RA.
Sponsor: Genentech, Inc. (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT3985g; WA20494
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Rheumatoid Arthritis
Keywords: anti-CD20; stage; CD20; RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo × 2 IV + MTX (Placebo Comparator): Participants received two intravenous (IV) infusion matching placebo to ocrelizumab on Day 1 and Day 15. A repeat course was administered at Weeks 24 and 26. Methotrexate 7.5-25 milligram (mg) was administered weekly.
  Interventions: Drug: Methotrexate; Drug: Placebo
- Ocrelizumab 200 mg × 2 IV + MTX (Experimental): Participants received two IV infusion of ocrelizumab 200 mg on Day 1 and Day 15. A repeat course was administered at Weeks 24 and 26. Methotrexate 7.5-25 mg was administered weekly.
  Interventions: Drug: Methotrexate; Drug: ocrelizumab
- Ocrelizumab 500 mg × 2 IV + MTX (Placebo Comparator): Participants received two IV infusion of ocrelizumab 500 mg on Day 1 and Day 15. A repeat course was administered at Weeks 24 and 26. Methotrexate 7.5-25 mg was administered weekly.
  Interventions: Drug: Methotrexate; Drug: ocrelizumab

INTERVENTIONS:
Drug: Methotrexate — Methotrexate tablet was administered orally at a dose 7.5-25 mg
Drug: ocrelizumab — Ocrelizumab was administered via IV infusion at a dose specified in arm description
  Arms: Ocrelizumab 200 mg × 2 IV + MTX; Ocrelizumab 500 mg × 2 IV + MTX
Drug: Placebo — Matching placebo to ocrelizumab was administered via IV infusion
  Arms: Placebo × 2 IV + MTX

SUMMARY:
This study will evaluate the efficacy and safety of ocrelizumab, compared with placebo, in combination with methotrexate in patients with active rheumatoid arthritis who have had an inadequate response to methotrexate. Patients will be randomized to receive placebo, 200mg of intravenous ocrelizumab or 500mg of i.v. ocrelizumab on Days 1 and 15. A repeat course of i.v. treatment will be administered at Weeks 24 and 26. All patients will receive 7.5mg - 25mg/week concomitant methotrexate at a stable dose. The anticipated time on study treatment is 1-2 years. Target sample size is 1000.

ELIGIBILITY:
Inclusion criteria:

* Adult patients, ≥18 years of age
* Rheumatoid arthritis for ≥ 3 months
* Inadequate clinical response to methotrexate at a dose of 7.5-25mg/week for ≥ 12 weeks

Exclusion criteria:

* Rheumatic autoimmune disease or inflammatory joint disease, other than RA
* Prior receipt of any biologic therapy for RA
* Concurrent treatment with any DMARD (other than methotrexate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1015 (Actual)
Dates: Start 2006-12-27 (Actual); Primary Completion 2009-10-06 (Actual); Study Completion 2015-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Dummer, M.D., Study Director — Genentech, Inc.
Locations (1):
- Trial Information Support Line, South San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Emery P, Rigby W, Tak PP, Dorner T, Olech E, Martin C, Millar L, Travers H, Fisheleva E. Safety with ocrelizumab in rheumatoid arthritis: results from the ocrelizumab phase III program. PLoS One. 2014 Feb 3;9(2):e87379. doi: 10.1371/journal.pone.0087379. eCollection 2014. PMID 24498318
- [Derived] Rigby W, Tony HP, Oelke K, Combe B, Laster A, von Muhlen CA, Fisheleva E, Martin C, Travers H, Dummer W. Safety and efficacy of ocrelizumab in patients with rheumatoid arthritis and an inadequate response to methotrexate: results of a forty-eight-week randomized, double-blind, placebo-controlled, parallel-group phase III trial. Arthritis Rheum. 2012 Feb;64(2):350-9. doi: 10.1002/art.33317. PMID 21905001

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Started | 324 | 344 | 347
Completed | 0 | 0 | 0
Not Completed | 324 | 344 | 347
Not completed — Death | 3 | 1 | 4
Not completed — Protocol Violation | 6 | 2 | 5
Not completed — Study Terminated by Sponsor | 260 | 288 | 282
Not completed — Withdrawal by Subject | 17 | 24 | 26
Not completed — Lack of Efficacy | 12 | 1 | 6
Not completed — Non-Compliance with Study Drug | 5 | 6 | 3
Not completed — Adverse Event | 10 | 12 | 16
Not completed — Lost to Follow-up | 11 | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX | Total
Number analyzed (Participants) | 320 | 343 | 343 | 1006
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.5 (11.54) | 51.8 (11.97) | 50.9 (12.23) | 51.1 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248 | 283 | 282 | 813
  Male | 72 | 60 | 61 | 193

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 20 Response at Week 24
Description: ACR20 is defined as 20 percent improvement respectively in: a) swollen joint count (SJC) and tender joint count (TJC) and b) Three of the following 5 assessments: Subject's global assessment of pain by VAS Subject's global assessment of disease activity (VAS) Investigator/Physician's global assessment of disease activity (VAS) Subject's assessment of disability measured by HAQ-DI Acute phase reactant (ESR or CRP).
Time Frame: Week 24
Population: ITT population included all randomised participants who had received any part of an infusion of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 320 | 343 | 343
Percentage of participants | 35.7 [30.5 to 41.0] | 56.9 [51.6 to 62.1] | 54.5 [49.2 to 59.8]
Statistical Analysis 1: Comparison: Placebo × 2 IV + MTX vs Ocrelizumab 200 mg × 2 IV + MTX; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted difference = 18.5, 95% CI 2-sided [11 to 25.9]
Statistical Analysis 2: Comparison: Placebo × 2 IV + MTX vs Ocrelizumab 500 mg × 2 IV + MTX; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted difference = 21.4, 95% CI 2-sided [14.1 to 28.8]

2. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 20 Response at Week 48
Description: as for outcome 1
Time Frame: Week 48
Population: ITT population included all randomised participants who had received any part of an infusion of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 320 | 343 | 343
Percentage of participants | 27.6 [22.7 to 32.5] | 58.3 [53.1 to 63.5] | 62.1 [57.0 to 67.2]
Statistical Analysis 1: Comparison: Placebo × 2 IV + MTX vs Ocrelizumab 200 mg × 2 IV + MTX; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted difference = 30.8, 95% CI 2-sided [23.7 to 37.9]
Statistical Analysis 2: Comparison: Placebo × 2 IV + MTX vs Ocrelizumab 500 mg × 2 IV + MTX; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted difference = 34.5, 95% CI 2-sided [27.4 to 41.5]

3. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a subject administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. Pre-existing conditions which worsened during the study were also reported as AEs.
Time Frame: From baseline up to 8.5 years
Population: The safety population included all participants who were randomized and received any part of an infusion of study drug and provided at least one assessment of safety.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 320 | 343 | 343
Percentage of participants | 79.4 | 82.2 | 83.7

4. Secondary Outcome: Percentage of Participants With a Major Clinical Response (ACR70 for ≥ 6 Months) at Week 48
Description: ACR70 is defined as 70 percent improvement respectively in: a) swollen joint count (SJC) and tender joint count (TJC) and b) Three of the following 5 assessments: Subject's global assessment of pain by VAS Subject's global assessment of disease activity (VAS) Investigator/Physician's global assessment of disease activity (VAS) Subject's assessment of disability measured by HAQ-DI Acute phase reactant (ESR or CRP).
Time Frame: Week 48
Population: ITT population included all randomised participants who had received any part of an infusion of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 320 | 343 | 343
Percentage of participants | 0.9 [0.0 to 2.0] | 6.1 [3.6 to 8.7] | 7.3 [4.5 to 10.0]

5. Secondary Outcome: Percentage of Participants Achieving Disease Activity Score 28 (DAS28) Remission (DAS28 < 2.6) at Weeks 24 and 48
Description: The Disease Activity Score (DAS28) score is a measure of the subject's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity and Erythrocyte Sedimentation Rate (ESR). DAS28 total scores range from 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from Baseline indicated improvement.
Time Frame: Weeks 24 and 48
Population: ITT population included all randomised participants who had received any part of an infusion of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 319 | 343 | 343
Percentage of participants
  Week 24 | 5.3 [2.9 to 7.8] | 7.9 [5.0 to 10.7] | 10.8 [7.5 to 14.1]
  Week 48 | 5.3 [2.9 to 7.8] | 16.0 [12.2 to 19.9] | 17.5 [13.5 to 21.5]

6. Secondary Outcome: Change From Baseline in DAS28 at Weeks 24 and 48
Description: as for outcome 5
Time Frame: Weeks 24 and 48
Population: ITT population included all randomised participants who had received any part of an infusion of study medication.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 316 | 340 | 336
Units on a Scale
  Baseline | 6.42 (1.103) | 6.40 (1.143) | 6.40 (1.077)
  Change at Week: number analyzed (Participants) | 227 | 299 | 300
  Change at Week | -1.33 (1.329) | -2.00 (1.248) | -2.02 (1.310)
  Change at Week 48: number analyzed (Participants) | 187 | 271 | 278
  Change at Week 48 | -1.38 (1.290) | -2.42 (1.504) | -2.68 (1.475)

7. Secondary Outcome: European League Against Rheumatism (EULAR) Response Rates (Categorical DAS Responders) at Weeks 24 and 48
Description: DAS 28 score is a measure of the subject's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity and ESR. DAS28 total scores range from 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from Baseline indicated improvement. EULAR Good response: DAS28 ≤ 3.2 and a change from Baseline < -1.2. EULAR Moderate response: DAS28 >3.2 to ≤ 5.1 or a change from Baseline < -0.6 to ≥ -1.2.
Time Frame: Weeks 24 and 48
Population: ITT population included all randomised participants who had received any part of an infusion of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 320 | 343 | 343
Percentage of participants
  Week 24 | 41.6 | 68.8 | 70.0
  Week 48 | 35.3 | 65.9 | 72.0

8. Secondary Outcome: Percentage of Participants Achieving an ACR50 Response at Weeks 24 and 48
Description: ACR50 is defined as 50 percent improvement respectively in: a) swollen joint count (SJC) and tender joint count (TJC) and b) Three of the following 5 assessments: Subject's global assessment of pain by VAS Subject's global assessment of disease activity (VAS) Investigator/Physician's global assessment of disease activity (VAS) Subject's assessment of disability measured by HAQ-DI Acute phase reactant (ESR or CRP).
Time Frame: Weeks 24 and 48
Population: ITT population included all randomised participants who had received any part of an infusion of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 319 | 343 | 343
Percentage of participants
  Week 24 | 16.3 [12.2 to 20.4] | 31.8 [26.9 to 36.7] | 31.2 [26.3 to 36.1]
  Week 48 | 12.9 [9.2 to 16.5] | 39.9 [34.8 to 45.1] | 36.7 [31.6 to 41.8]

9. Secondary Outcome: Percentage of Participants Achieving an ACR70 Response at Weeks 24 and 48
Description: as for outcome 4
Time Frame: Weeks 24 and 48
Population: ITT population included all randomised participants who had received any part of an infusion of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 319 | 343 | 343
Percentage of participants
  Week 24 | 5.6 [3.1 to 8.2] | 14.3 [10.6 to 18.0] | 12.2 [8.8 to 15.7]
  Week 48 | 6.6 [3.8 to 9.3] | 20.7 [16.4 to 25.0] | 22.4 [18.0 to 26.9]

10. Secondary Outcome: Percent Change From Baseline in Swollen Joint Count (SJC) at Weeks 24 and 48
Description: 66 joints were assessed for swelling and joints are classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 66.
Time Frame: Baseline, Week 24, 48
Population: ITT population included all randomised participants who had received any part of an infusion of study medication.
Measure: Mean (Standard Deviation); unit: Percentage of Change
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 235 | 311 | 308
Percentage of Change
  Change at Week 24 | -38.20 (66.127) | -51.82 (80.805) | -54.76 (39.896)
  Change at Week 48: number analyzed (Participants) | 211 | 296 | 299
  Change at Week 48 | -39.39 (59.184) | -61.36 (44.414) | -64.22 (65.234)

11. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC) at Weeks 24 and 48
Description: 68 joints were assessed for tenderness and joints were classified as tender/not tender giving a total possible tender joint count score of 0 to 68.
Time Frame: Baseline, Weeks 24, 48
Population: ITT population included all randomised participants who had received any part of an infusion of study medication.
Measure: Mean (Standard Deviation); unit: Tendor joins
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 235 | 311 | 308
Tendor joins
  Change at Week 24 | -36.97 (58.675) | -55.11 (37.962) | -51.07 (49.700)
  Change at Week 48: number analyzed (Participants) | 211 | 296 | 299
  Change at Week 48 | -35.91 (64.358) | -61.51 (37.229) | -59.55 (48.474)

12. Secondary Outcome: Change From Baseline in Patient's Pain Visual Analogue Scale (VAS) at Weeks 24 and 48
Description: The patient assessed their pain on a 0 to 100 millimeters (mm) horizontal visual analogue scale (VAS). The left-hand extreme of the line equals 0 mm, and is described as "no pain" and the right-hand extreme equals 100 mm as "unbearable pain". A negative change indicated improvement.
Time Frame: Baseline, Week 24, 48
Population: ITT population included all randomised participants who had received any part of an infusion of study medication.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 230 | 307 | 304
Units on scale
  Change at Week 24 | -9.10 (109.646) | -32.02 (88.637) | -27.73 (139.732)
  Change at Week 48: number analyzed (Participants) | 206 | 293 | 295
  Change at Week 48 | -2.28 (148.933) | -38.86 (104.267) | -32.47 (197.692)

13. Secondary Outcome: Change From Baseline in Physician's Global VAS at Weeks 24 and 48
Description: The physician's global assessment of disease activity is assessed on a 0 to 100 millimetres (mm) horizontal visual analogue scale (VAS) by the physician. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm as "maximum disease activity" (maximum arthritis disease activity).
Time Frame: Baseline, Week 24, 48
Population: ITT population included all randomised participants who had received any part of an infusion of study medication.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 320 | 343 | 343
Units on scale
  Change at Week 24 | -40.23 (39.655) | -51.44 (34.669) | -53.02 (34.479)
  Change at Week 48 | -41.60 (43.285) | -61.29 (31.543) | -62.10 (30.866)

14. Secondary Outcome: Change From Baseline in Patient's Global VAS at Weeks 24 and 48
Description: The patient's global assessment of disease activity is assessed on a 0 to 100 millimeters (mm) horizontal visual analogue scale (VAS) by the patient. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 24, 48
Population: ITT population included all randomised participants who had received any part of an infusion of study medication.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 231 | 308 | 303
Units on scale
  Change at Week 24 | -20.73 (74.480) | -37.96 (83.908) | -36.99 (79.130)
  Change at Week 48: number analyzed (Participants) | 207 | 294 | 294
  Change at Week 48 | -17.13 (100.706) | -42.02 (103.526) | -55.26 (37.873)

15. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) at Weeks 24 and 48
Description: The serum concentration of C-Reactive Protein (CRP) is measured in milligrams per deciliter (mg/dL). A reduction in the level is considered an improvement.
Time Frame: Baseline, Week 24, 48
Population: ITT population included all randomised participants who had received any part of an infusion of study medication.
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 235 | 311 | 308
Milligrams per deciliter (mg/dL)
  Change at Week 24 | 11.64 (116.697) | -30.41 (109.193) | -23.07 (109.193)
  Change at Week 48: number analyzed (Participants) | 211 | 296 | 299
  Change at Week 48 | 22.01 (190.346) | -40.89 (90.139) | 15.14 (820.007)

16. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire Disability Index (HAQ-DI) at Weeks 24 and 48
Description: HAQ-DI is a self-completed patient questionnaire specific for Rheumatoid Arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities. Each domain has at least 2 component questions. There are 4 possible responses for each component 0=without any difficulty 1=with some difficulty 2=with much difficulty 3=unable to do. Calculate HAQ-DI the patient must have a domain score for at least 6 of 8 domains. The HAQ-DI is the sum of the scores, divided by the number of domains that have a score (in range 6-8) for a total possible score minimum/maximum 0 (best) to 3 (worst). A negative change from baseline indicated improvement.
Time Frame: Baseline, Week 24, 48
Population: ITT population included all randomised participants who had received any part of an infusion of study medication. Here, 'n' signifies the number of partcipants evaluated at a specified time point.
Measure: Mean (Standard Deviation); unit: Percentage Change from Baseline
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 320 | 343 | 343
Percentage Change from Baseline
  Change at Week 24 | -20.11 (48.921) | -30.12 (86.217) | -40.83 (38.243)
  Change at Week 48 | -22.67 (57.893) | -35.47 (78.670) | -45.63 (39.241)

17. Secondary Outcome: Change From Baseline in the Erythrocyte Sedimentation Rate (ESR) at Weeks 24 and 48
Description: as for outcome 16
Time Frame: Baseline, Week 24, 48
Population: ITT population included all randomised participants who had received any part of an infusion of study medication. Here, 'n' signifies the number of participants evaluated at a specified time point.
Measure: Mean (Standard Deviation); unit: Percentage Change from Baseline
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 234 | 311 | 308
Percentage Change from Baseline
  Change at Week 24 | -2.51 (66.453) | -20.10 (90.059) | -29.98 (57.195)
  Change at Week 48: number analyzed (Participants) | 211 | 296 | 299
  Change at Week 48 | -2.72 (57.893) | -27.24 (147.973) | -41.19 (55.485)

18. Secondary Outcome: Change From Baseline in the Modified Total Sharp Score (mTSS) at Weeks 24 and 48
Description: mTSS: measure of joint damage that combines scores for bone erosion and joint space narrowing (JNS). Erosion score: total of 14 locations in each hand and wrist and 6 joints in the foot were evaluated for erosion using an 8-point scale where 0=normal to 3.5=very severe erosion. JNS score: total of 13 locations in each hand and wrist and 6 joints in the foot were evaluated for joint narrowing score using a 9-point scale where 0=normal to 4.0=definite ankylosis (stiffness or fixation of a joint). mTSS scores ranged from 0 (normal) to 292 (worst possible total score). Change= mTSS score at Week 24 minus score at baseline. An increase in mTSS from baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement.
Time Frame: Baseline, Week 24, 48
Population: mITT population. Number of participants analysed signifies participants who were evaluated for the endpoint.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 305 | 322 | 320
Units on scale
  Baseline | 33.58 (51.106) | 31.45 (51.323) | 31.99 (49.602)
  Change at Week 24: number analyzed (Participants) | 268 | 308 | 313
  Change at Week 24 | 1.04 (2.842) | 0.34 (2.424) | -0.03 (2.534)
  Change at Week 48: number analyzed (Participants) | 268 | 308 | 313
  Change at Week 48 | 1.74 (5.293) | 0.26 (2.791) | -0.03 (2.911)

19. Secondary Outcome: Change From Baseline in Modified Erosion Score at Weeks 24 and 48
Description: The erosion score is a summary of erosion severity in 32 joints of the hands (16 joints per hand) and 12 joints in the feet (6 joints per foot). Each joint is scored, according to the surface area involved, from 0 to 5, with 5 indicating extensive loss of bone from more than one-half of the articulating bone (0 indicates no erosion). Because each side of a foot joint is graded separately on this scale, the maximum erosion score for a foot joint is 10. The maximal erosion score is 280.
Time Frame: Baseline, Week 24, 48
Population: mITT population included all participants who were in the ITT analysis set and had both baseline radiograph and at least one post-baseline radiograph for campaign 1. Here, the number of participants analysed signifies participants who were evaluated for the endpoint.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 305 | 322 | 329
Units on scale
  Baseline | 17.10 (27.256) | 16.22 (27.875) | 16.24 (26.103)
  Change at Week 24: number analyzed (Participants) | 268 | 308 | 313
  Change at Week 24 | 0.61 (1.778) | 0.18 (1.487) | 0.04 (1.511)
  Change at week 48: number analyzed (Participants) | 268 | 308 | 313
  Change at week 48 | 1.06 (3.238) | 0.08 (1.690) | -0.08 (1.588)

20. Secondary Outcome: Change From Baseline in Modified Joint Space Narrowing Score at Weeks 24 and 48
Description: The joint space narrowing score summarizes the severity of joint space narrowing in 30 joints of the hands and 12 joints of the feet. Assessment of joint space narrowing for each hand (15 joints per hand) and foot (6 joints per foot), including subluxation, is scored from 0 to 4, with 0 indicating no/normal joint space narrowing and 4 indicating complete loss of joint space, bony ankylosis, or luxation. The maximum joint space narrowing score is 168.
Time Frame: Baseline, Week 24, 48
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 305 | 322 | 329
Units on scale
  Baseline | 16.47 (25.990) | 15.22 (25.012) | 15.75 (25.118)
  Change at Week 24: number analyzed (Participants) | 268 | 308 | 313
  Change at Week 24 | 0.43 (1.654) | 0.16 (1.655) | -0.07 (1.504)
  Change at Week 48: number analyzed (Participants) | 268 | 308 | 313
  Change at Week 48 | 0.68 (2.777) | 0.18 (1.471) | 0.05 (1.859)

21. Secondary Outcome: Percentage of Participants Without Radiographic Progression Defined as Change in mTSS ≤ 0 at Weeks 24 and 48
Description: Radiographic progression was defined as a change of ≤ 0 in the total Genant-modified Sharp score. The Genant-modified Sharp scoring system assesses structural damage due to rheumatoid arthritis in radiographs. A score for erosions of 0-3.5 (8 gradations) is assigned for 14 joints in each hand and wrist, and 6 joints in each foot. Joint space narrowing scores of 0-4 (9 gradations) are assigned to 13 joints in each hand and 6 joints in each foot. The maximum erosion score is 40 x 3.5 = 140. The maximum joint space narrowing score is 38 x 4.0 = 152. Both the erosion and joint space narrowing scores are normalized to 145 and are added together for a maximum total Genant-modified Sharp score of 290; the minimum score is 0. A higher score indicates more damage.
Time Frame: Weeks 24, 48
Population: The modified Intent-to-Treat (mITT) population included all participants who were in the ITT analysis set and had both baseline radiograph and at least one post-baseline radiograph for campaign 1. Here, the number of participants analysed signifies subjects who were evaluated for the endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 305 | 322 | 329
Percentage of Participants
  Week 24 | 47.5 [41.9 to 53.1] | 58.7 [53.3 to 64.1] | 65.3 [60.2 to 70.5]
  Week 48 | 37.7 [32.3 to 43.1] | 58.7 [53.3 to 64.1] | 60.8 [55.5 to 66.1]

22. Secondary Outcome: Percentage of Participants With a Reduction in Modified Total Sharp Score (mTSS) From Baseline at Week 48
Description: as for outcome 18
Time Frame: Baseline, Week 48
Population: mITT population. Number of participants analysed signifies participants who were evaluated for the endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 305 | 322 | 329
Percentage of Participants | 11.8 [8.2 to 15.4] | 22.7 [18.1 to 27.2] | 29.8 [24.8 to 34.7]

23. Secondary Outcome: Percentage of Participants With a Reduction of Greater Than or Equal to 0.25 Units in the HAQ-DI Score at Weeks 24 and
Description: as for outcome 16
Time Frame: Week 24, 48
Population: ITT population included all randomised participants who had received any part of an infusion of study medication. Here, the number of participants analysed signifies participants evaluated for this endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 319 | 343 | 343
Percentage of Participants
  Week 24 | 42.3 [36.9 to 47.7] | 59.8 [54.6 to 65.0] | 66.5 [61.5 to 71.5]
  Week 48 | 34.8 [29.6 to 40.0] | 58.9 [53.7 to 64.1] | 65.9 [60.9 to 70.9]

24. Secondary Outcome: Change From Baseline in Short Form Health Survey (SF-36) Subscale and Summary Scores at Weeks 24 and 48
Description: The SF-36 is a questionnaire used to assess physical functioning and is made up of eight domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health. Transforming and standardizing these domains leads to the calculation of the Physical and Mental Component Summary measures. Scores ranging from 0 to 100, with 0=worst score (or quality of life) and 100=best score. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 24, 48
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 312 | 334 | 334
Units on scale
  Baseline: Mental Component Summary | 40.54 (12.282) | 39.99 (11.863) | 40.48 (12.822)
  Change at Week 24: Mental Component Summary: number analyzed (Participants) | 229 | 303 | 302
  Change at Week 24: Mental Component Summary | 4.38 (10.886) | 6.11 (10.082) | 5.80 (11.224)
  Change at Week 48: Mental Component Summary: number analyzed (Participants) | 206 | 290 | 292
  Change at Week 48: Mental Component Summary | 4.15 (10.326) | 6.36 (10.212) | 6.43 (11.795)
  Baseline: Physical Component Summary | 31.86 (7.387) | 32.24 (7.401) | 31.58 (8.039)
  Change at Week 24: Physical Component Summary: number analyzed (Participants) | 229 | 303 | 302
  Change at Week 24: Physical Component Summary | 5.29 (8.421) | 6.73 (8.385) | 7.71 (7.328)
  Change at Week 48: Physical Component Summary: number analyzed (Participants) | 206 | 290 | 292
  Change at Week 48: Physical Component Summary | 5.28 (8.373) | 8.38 (8.347) | 9.15 (8.389)

25. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F) Fatigue Assessment at Weeks 24 and 48
Description: The FACIT-Fatigue score was calculated according to a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the participants fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). Clinically relevant improvement is defined as a greater than or equal to (≥)5-point change from Baseline.
Time Frame: Baseline, Week 24, 48
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 317 | 340 | 340
Units on scale
  Baseline | 27.25 (10.821) | 26.87 (10.920) | 26.57 (11.194)
  Change at Week 24: number analyzed (Participants) | 235 | 309 | 308
  Change at Week 24 | 5.14 (9.864) | 7.18 (9.755) | 7.07 (10.269)
  Change at Week 48: number analyzed (Participants) | 211 | 296 | 298
  Change at Week 48 | 5.39 (10.054) | 8.01 (10.132) | 8.41 (10.682)

26. Secondary Outcome: Change From Baseline in Pain Quality and Impact of Pain on Daily Function Measured by the Brief Pain Inventory (BPI) Short Form at Weeks 24 and 48
Description: The modified BPI (short-form) is a short questionnaire to assess the severity of pain and the impact of pain on daily functions. The first two questions relate to average and current pain respectively and are assessed on a scale from 0 to 10, where 0 represents no pain, and 10 represents pain as bad as one can imagine. The degree to which pain has interfered with 7 different aspects is also rated on a scale from 0 to 10, where 0 represents that pain does not interfere and 10 that pain completely interferes.
Time Frame: Baseline, Week 24, 48
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
Number analyzed (Participants) | 316 | 340 | 335
Units on scale
  Baseline: average pain | 6.39 (2.011) | 6.28 (2.077) | 6.42 (2.194)
  Baseline: pain right now | 5.57 (2.398) | 5.75 (2.495) | 5.82 (2.533)
  Change at Week 24: average pain: number analyzed (Participants) | 234 | 304 | 298
  Change at Week 24: average pain | -1.82 (2.441) | -2.45 (2.299) | -2.48 (2.424)
  Change at Week 24: pain right now: number analyzed (Participants) | 235 | 303 | 299
  Change at Week 24: pain right now | -1.57 (2.775) | -2.32 (2.659) | -2.24 (2.671)
  Change at Week 48: average pain: number analyzed (Participants) | 188 | 273 | 280
  Change at Week 48: average pain | -1.78 (2.619) | -2.92 (2.442) | -3.06 (2.422)
  Change at Week 48: pain right now: number analyzed (Participants) | 188 | 272 | 282
  Change at Week 48: pain right now | -1.53 (2.795) | -2.66 (2.676) | -2.92 (2.681)

ADVERSE EVENTS:
Time Frame: Baseline up to 33 months.
Description: All patients that received any part of an infusion of study drug and provided at least one assessment of safety were included in the safety population. In patients who had received the incorrect therapy from that intended were summarized in the group according to the highest dose of double-blind therapy they actually received.
Arm/Group | Placebo × 2 IV + MTX | Ocrelizumab 200 mg × 2 IV + MTX | Ocrelizumab 500 mg × 2 IV + MTX
All-Cause Mortality (participants affected / at risk) | 5/318 | 2/343 | 8/345
Serious Adverse Events (participants affected / at risk) | 73/318 | 61/343 | 78/345
Other Adverse Events (participants affected / at risk) | 228/318 | 272/343 | 273/345
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo × 2 IV + MTX (N=318) | Ocrelizumab 200 mg × 2 IV + MTX (N=343) | Ocrelizumab 500 mg × 2 IV + MTX (N=345)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vasculitis necrotising (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (3)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Inflammatory carcinoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Myxoid liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Drug dependence (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hypomania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Otosalpingitis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 3 (3) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Stag horn calculus (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urogenital fistula (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Basedow's disease (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (4) | 4 (4) | 10 (10)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (1) | 3 (3)
Cellulitis (Infections and infestations) | 3 (3) | 1 (1) | 3 (4)
Sepsis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Abscess soft tissue (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute hepatitis B (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Borrelia infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis gangrenous (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fungal oesophagitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
Histoplasmosis (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mycobacterium kansasii infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Purulent synovitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo × 2 IV + MTX (N=318) | Ocrelizumab 200 mg × 2 IV + MTX (N=343) | Ocrelizumab 500 mg × 2 IV + MTX (N=345)
Hypertension (Vascular disorders) | 26 (28) | 42 (43) | 37 (45)
Infusion related reaction (Injury, poisoning and procedural complications) | 62 (136) | 89 (164) | 96 (168)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 13 (15) | 20 (23)
Anaemia (Blood and lymphatic system disorders) | 17 (19) | 13 (14) | 13 (15)
Headache (Nervous system disorders) | 24 (29) | 29 (33) | 32 (38)
Oedema peripheral (General disorders) | 17 (21) | 16 (18) | 14 (15)
Depression (Psychiatric disorders) | 19 (19) | 18 (20) | 21 (23)
Insomnia (Psychiatric disorders) | 19 (19) | 19 (19) | 15 (16)
Diarrhoea (Gastrointestinal disorders) | 23 (28) | 21 (22) | 23 (29)
Dyspepsia (Gastrointestinal disorders) | 14 (15) | 17 (18) | 22 (24)
Gastritis (Gastrointestinal disorders) | 8 (9) | 14 (16) | 18 (18)
Nausea (Gastrointestinal disorders) | 17 (21) | 15 (17) | 22 (26)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (17) | 19 (20) | 26 (27)
Bronchitis (Infections and infestations) | 39 (57) | 43 (59) | 40 (47)
Gastroenteritis (Infections and infestations) | 16 (22) | 11 (12) | 15 (20)
Influenza (Infections and infestations) | 20 (26) | 31 (37) | 29 (35)
Herpes zoster (Infections and infestations) | 16 (17) | 14 (16) | 12 (13)
Nasopharyngitis (Infections and infestations) | 45 (60) | 43 (56) | 51 (77)
Pharyngitis (Infections and infestations) | 18 (22) | 9 (14) | 9 (13)
Sinusitis (Infections and infestations) | 18 (27) | 33 (48) | 28 (35)
Upper respiratory tract infection (Infections and infestations) | 64 (130) | 79 (130) | 85 (157)
Urinary tract infection (Infections and infestations) | 40 (67) | 38 (49) | 48 (69)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.